CLINICAL TRIAL: NCT03102021
Title: The Effect of High Dose Erythropoietin in Acute Renal Failure
Brief Title: The Effect of Human Recombinant Erythropoietin in Acute Renal Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Devasmita Dev, MD, Principal Investigator, North Texas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #05-141; 092006-064 - UTSW protocol ID
Record Dates: First submitted 2007-12-26; First posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Erythropoietin; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Active Comparator): erythropoeitin
  Interventions: Drug: erythropoietin
- 2 (Placebo Comparator): saline placebo
  Interventions: Drug: saline

INTERVENTIONS:
Drug: erythropoietin — 500 units/kg daily for 3 days at onset of acute kidney injury
  Other Names: erythropoeitin
  Arms: 1
Drug: saline — saline 10 ml for 3 days
  Other Names: normal saline
  Arms: 2

SUMMARY:
The purpose of this study is to determine if the use of erythropoietin when used in high dose during acute kidney injury can decrease the number of days of kidney injury.

DETAILED DESCRIPTION:
Acute kidney injury is associated with increased morbidity. The most common injury to the kidney occurs during hospitalization with either ischemic or nephrotoxic insult to the kidney. This can prolong hospitalization and depending on the severity of the insult result in permanent decreased kidney function. Recent studies in animals have suggested benefits of using erythropoietin in high doses at time of kidney injury with eividence for less injury in the kidney tissue of those animals who received treatment compared to those animals that received only saline. Limited human data also suggests that use of high dose erythropoietin at the time of stroke can decrease the extent of brain injury. In addition cardiac cell culture studies also have shown decrease in cell injury with use of erythropoietin. These studies have prompted us to evaluate if admininstering erythropoietin to those with onset of acute kidney injury during their hospitalization may benefit from this intervention. This pilot study then evaluates that use of high dose erythropoietin administed daily over 3 days in patients with acute kidney injury on whether the days spent in renal failure are less than those who will receive no study medication. Those patients with kidney failure from either ischemic or nephrotoxic insult and no other contraindication to erythropoietin use will be considered for the study. Informed consent is obtained from the patient or next of kin

ELIGIBILITY:
Inclusion Criteria:

* age equal or greater than 21 yo
* acute neprhotoxic or ischemic kidney injury, acute tubular necrosis

Exclusion Criteria:

* no active or current malignancies
* not actively receiveing epo
* GFR less than 60 ml/min
* unable to provide informed consent
* contraindication to erythropoietin use

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
days of acute renal failure | 28 days

SECONDARY OUTCOMES:
days of hospitalization | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Devasmita Dev, MD, Principal Investigator — DAllas VA Medical Center/UT Southwestern Medical Center
Locations (1):
- Dallas VAMC, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No